CLINICAL TRIAL: NCT00670579
Title: A Prospective Study About Complications of Totally Implantable Central Venous Access Ports in People With CF
Brief Title: Study About Complications of Totally Implanted Venous Access Devices (TIVADs) in People With Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Filippo Festini, Associate Professor, University of Florence
Other Study IDs: FFC#30/2008
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Cystic Fibrosis
Keywords: TIVAD; complications; nursing; cystic fibrosis; implanted
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pulmonary infections are the major cause of mortality and morbidity in cystic fibrosis (CF); patients frequently have to take antibiotics which often cannot be given orally or by aerosol but have to be administered intravenously. In order to reduce the number of venepunctures, totally implanted venous access devices (TIVAD) or Ports have been used to administer antibiotics and other infusions.

The use of Port systems has been increasing in recent years, especially for those patients requiring frequent intravenous treatments. Having a TIVAD in place makes venous access quicker and also reduces trauma, suffering and pain. However, there are important complications associated with TIVADs which can be early (pneumothorax, arterial puncture, severe bruising) or late (infections, thromboembolic complications and occlusion).

Although the use of TIVADs in CF is increasing, there is little CF-specific literature available on the epidemiology and risk of TIVAD complications. Also, literature is scarce about clinical criteria for deciding to insert a TIVAD. Therefore, so far clinical decisions were based mainly on experiences of TIVAD use in other diseases, such as cancer.

With this prospective observational study we will survey a large population of Italian CF people with TIVAD in order to: collect data about current clinical conditions of CF people with TIVAD; investigate about clinical criteria that led to the decision of positioning a TIVAD; observe the possible onset of late complications.

DETAILED DESCRIPTION:
To be included in the study, subjects need to fulfil the following requirements:

* Diagnosis of CF, made accordingly to the CF Foundation Guideline;
* Ability to consciously express owns informed consent, if aged 18 or more. If minor, presence of at least one legally authorised parent able to consciously express informed consent;
* Have a TIVAD implanted;
* Have no current complications in the TIVAD (infection, thromboembolic complications or occlusion) Outcome Measures

Measured outcomes will be:

1. Incidence of TIVAD infections (Port pocket infection, Cutaneous site infection,Catheter-related infection;
2. Incidence of TIVAD thrombosis;
3. Incidence of TIVAD occlusion.

The observational phase will last 12 months for each subject involved

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF, made accordingly to the CF Foundation Guideline
* Ability to consciously express owns informed consent, if aged 18 or more. If minor, presence of at least one legally authorised parent able to consciously express informed consent
* Have a TIVAD implanted
* Have no current complications in the TIVAD (infection, thromboembolic complications or occlusion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with CF and with a TIVAD implanted
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of late complications (infectious, thrombotic and obstructive) in CF people with a totally implanted venous access devices and to investigate possible associations between the onset of complications and several variables | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cystic Fibrosis Center of Tuscany, Meyer Hospital, Florence, Tuscany, Italy